CLINICAL TRIAL: NCT04438928
Title: Effects of Multiple Micronutrients and Docosahexaenoic Acid (DHA) Supplementation During Pregnancy on Maternal Biomarkers and Infant Anthropometric Outcomes
Brief Title: Clinical Study on the Effect of Elevit Pregnancy 2nd & 3rd Trimester (Multi-micronutrients & DHA Supplement) on the Nutritional Status of Pregnant Women During Second and Third Trimester
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 18366
Record Dates: First submitted 2020-05-29; First posted 2020-06-19 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Healthy Pregnant Women
MeSH Terms: interventions — Pregnancy Trimester, Third

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy pregnant women - Supplement (Experimental): Supplementation with micronutrients plus docosahexaenoic acid (DHA) preparation (Multimicronutrients and docosahexaenoic acid (MMS) soft gel capsules) during 2nd and 3rd trimesters of pregnancy.
  Subgroup: Healthy pregnant women with Caesarean section [A subset of subjects (approximately 10 subjects per study arm) undergoing elective Caesarean section (for reasons independent from the study)]
  Interventions: Dietary Supplement: Elevit Pregnancy 2nd & 3rd Trimester
- Healthy pregnant women - Non-Supplement (Other): Control study group
  Subgroup: Healthy pregnant women with Caesarean section [A subset of subjects (approximately 10 subjects per study arm) undergoing elective Caesarean section (for reasons independent from the study)]
  Interventions: Other: Non-Supplement

INTERVENTIONS:
Dietary Supplement: Elevit Pregnancy 2nd & 3rd Trimester — Once daily micronutrient plus DHA supplementation (Multi-micronutrients and docosahexaenoic acid (MMS) soft gel capsules)
  Other Names: BAY 987765 Multi-micronutrient & DHA
  Arms: Healthy pregnant women - Supplement
Other: Non-Supplement — Control study group of pregnant women non-supplemented with multi-micronutrients and docosahexaenoic acid (MMS) soft gel capsules
  Arms: Healthy pregnant women - Non-Supplement

SUMMARY:
The aim of this study is to collect information how adding a soft gel preparation of micronutrients such as vitamins, dietary minerals plus omega-3 fatty acid (docosahexaenoic acid, DHA) to the diet of pregnant women during the 2nd and 3rd trimesters of pregnancy effects the nutritional state of the mother and infants at delivery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant Caucasian women aged 18 to 42 years (inclusive) in their 1st - 2nd trimester (gestational age (GA) week 11-14 at screening);
* Hemoglobin (Hg) > 105g/L;
* Inconspicuous fetal anomaly screening;
* Normal ultrasound examination (Ultra Sonography (USG));
* Singleton pregnancy;
* Taking at least 400 mcg folate per day;
* Seronegative for Human Immunodeficiency Virus (HIV), Hepatitis B and Hepatitis C at screening;
* Pregnant women who, in the opinion of the Investigator, are willing and able to participate in all scheduled visits, to adhere to the supplementation plan, to laboratory tests and to all other study related procedures according to the clinical protocol;
* Pregnant women providing a personally signed and dated given informed consent to participate in the study and to adhere to all study procedures indicating that they have been informed of all pertinent aspects of the trial and that they understood and accepted these, prior to admission to the study.

Exclusion Criteria:

* Physical (including vital signs e.g. blood pressure and pulse rate), hematological and clinical-chemical parameters deviating from normal and with clinical relevance;
* Any infection (acute or chronic) at screening and baseline;
* Any current metabolic diseases (e.g. diabetes, hypothyroidism);
* Less than 12 months from previous delivery;
* Any history or current diseases, which are associated with malabsorption, or other severe diseases of the gastrointestinal tract (e.g. chronic inflammatory bowel disease, iron accumulation, iron utilization disorders); Any history or current neurological, cardiac, endocrine or bleeding disorders;
* Specific diets (e.g. vegan vegetarian, celiac, lactose free);
* Body mass index (BMI) < 18 or >30 kg/m2;
* Pregnant women already taking DHA/multivitamin supplements (except folate or iron);
* Diagnosed or suspected malignant or premalignant disease;
* Current clinically significant depression;
* Current intake of pharmaceuticals or dietary supplements which may interact with any of the ingredients of the trial treatment (i.e. fluoroquinolones, bisphosphonates, levodopa, levothyroxine, penicillamine, antibiotics containing tetracycline or trietine);
* History of or current diseases where vitamin, mineral, trace element or DHA supplementation might be not recommended /contraindicated [such as sickle cell anemia, copper metabolism disorders (Wilson's disease), renal disease, nephrolithiasis, urolithiasis, hypercalcemia, hypercalciuria, hepatobiliary diseases, existing hypervitaminosis, iron metabolism disorders, hypermagnesemia];
* Severe Hyperemesis gravidarum;
* Previous adverse birth outcomes (e.g. small for gestational age, low birth weight, premature birth, stillbirth, more than two consecutive spontaneous abortions);
* Previous adverse pregnancy outcomes (e.g. gestational diabetes);
* Diagnosed congenital abnormalities in current or previous pregnancy;
* Known carrier or affected with a genetic disease or condition (e.g. mutation carrier for autosomal recessive diseases);
* History of or current abuse of drugs, alcohol or other substances;
* Current smokers and women who smoked during current pregnancy;
* Any history of hypersensitivity or known allergy to any of the ingredients of the study supplement.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 164 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline: Blood RBC DHA/wt% TFA | Baseline: Screening at gestational age (GA) week 11 to 13 and at GA week 24 to 26 and week 34 to 36
  In order to assess the beneficial effects of supplementation with micronutrients and DHA (docosahexaenoic acid) during 2nd and 3rd trimesters of pregnancy, the red blood cell (RBC) DHA weight percent of total fatty acids (DHA wt% TFA) will be measured compared to baseline as primary maternal variable.
  Gestational age is a measure of the age of a pregnancy which is taken from the beginning of the woman's last menstrual period (LMP), or the corresponding age of the gestation as estimated by a more accurate method if available. Such methods include adding 14 days to a known duration since fertilization (as is possible in in vitro fertilization), or by obstetric ultrasonography. The popularity of using such a definition of gestational age is that menstrual periods are essentially always noticed, while there is usually a lack of a convenient way to discern when fertilization occurred.

SECONDARY OUTCOMES:
Change from baseline: Blood RBC EPA/wt% TFA | Baseline: Screening at gestational age (GA) week 11 to 13 and at GA week 24 to 26 and week 34 to 36
  Red blood cell (RBC) EPA (eicosapentaenoic acid) weight percent of total fatty acids (DHA wt% TFA).
Change from baseline: Blood RBC DHA/TFA ratio % | Baseline: Screening at gestational age (GA) week 11 to 13 and at GA week 24 to 26 and week 34 to 36
Change from baseline: Blood RBC Omega 3 index in RBC | Baseline: Screening at gestational age (GA) week 11 to 13 and at GA week 24 to 26 and week 34 to 36
  The "omega-3 index" reflects the content of EPA plus DHA in erythrocyte membranes expressed as a percentage of total erythrocyte fatty acids.
Change from baseline: Blood 25-hydroxyvitamin D concentration % | Baseline: Screening at gestational age (GA) week 11 to 13 and at GA week 24 to 26 and week 34 to 36
Change from baseline: Blood Glutathione (GSH)/oxidized Glutathione (GSSG) ratio % | Baseline: Screening at gestational age (GA) week 11 to 13 and at GA week 24 to 26 and week 34 to 36
  Glutathione exists in reduced (GSH) and oxidized (GSSG) states. Reduced glutathione is the most abundant antioxidant in aerobic cells and participates in the detoxification of lipid hydroperoxides and hydrogen peroxide exerted by glutathione peroxidases. When cells are exposes to increased oxidative stress levels, GSSG accumulates and the GSH/GSSG ratio decreases.
Change from baseline: Blood Reactive oxygen metabolites (ROMs) concentrations % | Baseline: Screening at gestational age (GA) week 11 to 13 and at GA week 24 to 26 and week 34 to 36
Change from baseline: Blood 8-Isoprostane concentration % | Baseline: Screening at gestational age (GA) week 11 to 13 and at GA week 24 to 26 and week 34 to 36
Infant sex | At delivery
Infant gestational age | At delivery
Infant head circumference | At delivery
Infant weight measurements | At delivery
Infant length measurements | At delivery
Infant ponderal index | At delivery
Infant skinfold thickness | At delivery
  Triplicate measurements: triceps, biceps, suprailiac, and subscapular on left side with standard skinfold caliper operated with constant pressure of 10 g/mm2)
Infant Apgar score | At delivery
Infant bone density | Up to 10 days after delivery
Umbilical cord blood gas analysis | At delivery
  Cord blood sample evaluations in a subset of women undergoing Caesarean section.
Umbilical cord blood pH analysis | At delivery
  Cord blood sample evaluations in a subset of women undergoing Caesarean section.
Cord blood metabolomic analysis | At delivery
  Cord blood sample evaluations in a subset of women undergoing Caesarean section.
Placental weight | At delivery
  Placenta tissue sample evaluation in a subset of women undergoing caesarean section.
  Placental efficiency will be estimated through the feto/placental weight (F/P) ratio, calculated as birth weight divided by the placental weight.
Placental biometric parameters | At delivery
  Placenta tissue sample evaluation in a subset of women undergoing caesarean section.
  i.e. larger (D) and smaller (d) diameters of the chorionic elliptical disc, feto/placental weight (F/P ratio)
Blood, cord blood and placental RBC DHA/wt% TFA | At delivery
  Sample evaluations in a subset of women undergoing Caesarean section.
Blood, cord blood and placental RBC EPA wt% TFA | At delivery
  Sample evaluations in a subset of women undergoing Caesarean section.
Blood, cord blood and placental DHA/TFA ratio % | At delivery
  Sample evaluations in a subset of women undergoing Caesarean section.
Blood, cord blood and placental RBC Omega 3 index | At delivery
  Sample evaluations in a subset of women undergoing Caesarean section.
Mitochondrial DNA content evaluation in placental tissue and isolated trophoblast cells | At delivery
  mtDNA is a well-accepted molecular marker to assess mitochondria content.
  Sample evaluations in a subset of women undergoing Caesarean section.
IL-6 (Interleukin 6), IL-10 (Interleukin 10) and TNF-α (Tumor Necrosis Factor Alpha) in placental tissue and isolated trophoblast cells | At delivery
  These genes are constitutively expressed in human placenta and are a reliable marker of inflammation.
  Sample evaluations in a subset of women undergoing Caesarean section.
Placental tissue metabolomic analysis | At delivery
  Sample evaluations in a subset of women undergoing Caesarean section.
  The rationale for conducting metabolomic analysis is to understand if multi-micronutrient supplement (MMS) supplementation during the second and third trimester of pregnancy influences maternal and infant gestational outcomes (e.g. oxidative stress, placental function).
Blood, cord blood and placental 8-isoprostane | At delivery
  Sample evaluations in a subset of women undergoing Caesarean section.
Blood, cord blood and placental reactive oxygen metabolites (ROMs) concentrations % | At delivery
  Sample evaluations in a subset of women undergoing Caesarean section.
Number of Adverse Events (AEs) | Within 7 days after Delivery
Severity of AEs | Within 7 days after Delivery
AE relationship to the investigational product | Within 7 days after Delivery

OTHER OUTCOMES:
Maternal Food Frequency Questionnaire FFQ | Up to GA week 34-36
  Focus on foods providing DHA

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- ASST Fatebenefratelli Sacco, Milan, Lombardy, Italy

REFERENCES:
- [Derived] Parisi F, Mando C, Novielli C, Anelli GM, Cazzola R, Lisso F, Sarno L, Marelli E, Lubrano C, Maria Antonazzo PG, Cetin I. Maternal mid-pregnancy long-chain polyunsaturated fatty acid profile is associated with pregestational body mass index and neonatal anthropometric measures at birth among non-obese pregnancies: results from two Italian multicenter cohorts. Nutr Metab (Lond). 2025 Nov 12;22(1):137. doi: 10.1186/s12986-025-01034-8. PMID 41225593